CLINICAL TRIAL: NCT02427126
Title: Apixaban for Treatment of Embolic Stroke of Undetermined Source (ATTICUS Randomized Trial)
Brief Title: Apixaban for Treatment of Embolic Stroke of Undetermined Source
Acronym: ATTICUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Bristol-Myers Squibb (Industry); Medtronic (Industry); ZKS and IKEaB Tübingen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-005109-19
Record Dates: First submitted 2015-03-20; First posted 2015-04-27 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: ESUS; anticoagulation
MeSH Terms: interventions — apixaban; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apixaban (Experimental): Apixaban 5mg b.i.d. Study treatment: 12 months Follow-up: 30 days after last study drug intake
  Interventions: Drug: Apixaban
- Aspirin (Active Comparator): Acetylic Salicylic Acid 100mg o.d.; Study treatment: 12 months Follow-up: 30 days after last study drug intake
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Apixaban — Apixaban is an oral anticoagulant currently approved for prevention of stroke and systemic embolism in patients with non-valvular atrial fibrillation, for the treatment of deep vein thrombosis and pulmonary embolism, and for the prophylaxis of systemic embolism after orthopedic surgery
  Other Names: Eliquis
  Arms: Apixaban
Drug: Aspirin — Acetylic Salicylic Acid 100mg o.d.; 12 Months
  Arms: Aspirin

SUMMARY:
Multicentre (national, Germany), randomized (2x2 factorial), open, parallel group, active controlled, efficacy study (phase III)

DETAILED DESCRIPTION:
Based on the previous data, ATTICUS is designed as multicentre, national, parallel group, active controlled, phase III randomized (2x2 factorial), clinical trial to demonstrate the superiority of apixaban against the current standard of treatment (acetylsalicylic acid) for the longterm treatment after ESUS. ATTICUS will follow a dynamic treatment protocol implementing conversion from the acetylsalicylic acid arm to the apixaban arm in case of detection of relevant episodes of AF during the course of the study. ATTICUS is designed to test the superiority over acetylsalicylic acid to reduce new ischemic lesion detected by FLAIR/DWI MRI.

ELIGIBILITY:
Inclusion criteria Must be ≥ 18 years at the time of signing the informed consent.

* ESUS must be defined according to following criteria:

  * Stroke detected by CT or MRI that is not lacunar
  * Absence of extracranial or intracranial atherosclerosis causing ≥50% luminal stenosis in arteries supplying the area of ischaemia
  * No major-risk cardioembolic source of embolism
  * No other specific cause of stroke identified
* * At least one of the following non-major but suggestive risk factors for cardiac embolism:

  * LA size >45mm (parasternal axis)
  * spontaneous echo contrast in LAA
  * LAA flow velocity <=0.2m/s
  * atrial high rate episodes
  * CHA2DS2-Vasc score >=4
  * persistent foramen ovale
* Understand and voluntarily sign an informed consent document
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception.

Exclusion Criteria:

* History of hypersensitivity to the investigational medicinal product
* Participation in other clinical trials or observation period of competing trials.
* Arteria cerebri media stroke affecting > 30% of c o r r e s p o n d i n g territory
* Diagnosis of haemorrhage or other pathology,
* Clear indication for anticoagulation
* Inability to control following risk factors for Hemorrhagic Transformation of fresh cerebral Infarction (HTI) during index hospital stay: presence of HTI at the time of anticoagulation, blood pressure >140 mmHg systolic, abnormal blood glucose Clear indication for dual antiplatelet therapy
* Clear stroke-/non-stroke-indication for concomitant long-term therapy with antiplatelets (e.g. acetylsalicylic acid (ASA), Clopidogrel, or Prasugrel) or with non-steroidal anti-inflammatory drugs (NSAID).
* Concomitant systemic therapy with strong inhibitors of cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp), i.e. azole antimycotics and human immunodeficiency virus (HIV)-protease inhibitors.
* Contraindication to investigational medications
* Planned or likely therapy with fibrinolytic agents within 48 hours of first study medication
* History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
* Gastrointestinal bleed or major surgery within 3 months
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
* TIA or minor stroke induced by angiography or surgery
* Severe non-cardiovascular comorbidity with life expectancy < 3 months
* Severe renal failure, defined as Glomerular Filtration Rate (GFR) <15ml/min
* Severe hepatic insufficiency (Child-Pugh score B to C),
* Active liver disease,
* Contraindications against performance of MRI (pacemaker/ICD), previous implantation non-MRI capable protheses
* Patients considered unreliable by the investigator, or having a life expectancy less than the expected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Imaging Endpoint: Occurrence of at least one new ischemic lesion at 12 months after study drug initiation when compared to baseline MRI before study drug initiation | 12 months
  The primary endpoint will be the occurrence of at least one new ischemic lesion identified by magnetic resonance imaging (axial T2-weighted fluid attenuated inversion recovery MRI (FLAIR) and/or axial diffusion weighted MRI (DWI)) at 12 months when compared to the baseline MRI (FLAIR, DWI) obtained at the time of study drug initiation. MRI at 12 months will be directly compared with the baseline MRI to assess for new ischemic lesions.

SECONDARY OUTCOMES:
Combination of recurrent ischaemic stroke, hemorrhagic stroke, systemic embolism | 12 months
  The occurence of ischaemic stroke, hemorrhagic stroke, or systemic embolism during study participation (12months) will be quantified
Combination of major adverse cardiovascular events (MACE) including recurrent stroke, myocardial infarction and cardiovascular death | 12 months
  The occurence of major adverse cardiovascular events (MACE) including recurrent stroke, myocardial infarction and cardiovascular death during study participation (12months) will be quantified
Combination of major and clinically relevant non-major bleedings defined according to ISTH criteria | 12 months
  The occurence of major and clinically relevant non-major bleedings defined according to ISTH criteria during study participation (12months) will be quantified
Change of cognitive function (MOCA) | 12 months
  MOCA test will be performed upon study enrollment and 12 months after enrollment and both tests will be compared
Life quality (EQ-5D) | 12 months
  EQ-5D questionnaire will be raised upon study enrollment and 12 months after enrollment and both questionnaires will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Geisler, Prof, Principal Investigator — Tübingen University Hospital; Sven Poli, Prof, Principal Investigator — Tübingen University Hospital; Schreieck Jürgen, Prof, Principal Investigator — Tübingen University Hospital
Locations (16):
- Germany (16):
  - MedicalPark Berlin Humboldtmühle GmbH & Co. KG, Berlin
  - Neurologische Klinik, Universität Bonn, Bonn
  - Regiomed Kliniken Coburg GmbH Abt. II, Coburg
  - Neurologie, Klinikum Friedrichshafen GmbH, Friedrichshafen
  - Universitätsmedizin Göttingen Abt.Innere Medizin, Klinik für Kardiologie und Pneumologie,, Göttingen
  - Krankenhaus Martha-Maria Halle-Döhlau, Halle
  - Klinik für Neurolgie,UKSH Campus Kiel, Kiel
  - Klinik für Neurologie, Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsklinik für Neurologie, Magdeburg, Magdeburg
  - Carl von Basedow KlinikumSaalekreis gGmbH, Merseburg
  - Marienhospital Stuttgart, Klinik für Neurologie, Stuttgart
  - Neurologische Klinik des Bürgerhospitals, Stuttgart
  - University Hospital, Tübingen
  - Universitäts- und Rehabilitationskliniken Ulm,Klinik für Neurologie, Ulm
  - Schwarzwald Baar Klinikum GmbH, Villingen-Schwenningen
  - Rems-Murr-Klinikum WinnendenNeurologie, Winnenden

REFERENCES:
- [Derived] Geisler T, Keller T, Martus P, Poli K, Serna-Higuita LM, Schreieck J, Gawaz M, Tunnerhoff J, Bombach P, Nagele T, Klose U, Aidery P, Groga-Bada P, Kraft A, Hoffmann F, Hobohm C, Naupold K, Niehaus L, Wolf M, Bazner H, Liman J, Wachter R, Kimmig H, Jung W, Huber R, Feurer R, Lindner A, Althaus K, Bode FJ, Petzold GC, Nguyen TN, Mac Grory B, Schrag M, Purrucker JC, Zuern CS, Ziemann U, Poli S; ATTICUS Investigators. Apixaban versus Aspirin for Embolic Stroke of Undetermined Source. NEJM Evid. 2024 Jan;3(1):EVIDoa2300235. doi: 10.1056/EVIDoa2300235. Epub 2023 Dec 22. PMID 38320511